CLINICAL TRIAL: NCT02602262
Title: Observational Study of HIV+ Deceased Donor Solid Organ Transplant for HIV+ Recipients
Brief Title: Observational Study of HIV+ Deceased Donor Transplant for HIV+ Recipients
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: University of Colorado, Denver (Other); Yale University (Other); Georgetown University (Other); Emory University (Other); Rush University Medical Center (Other); University of Illinois at Chicago (Other); Indiana University (Other); University of Maryland (Other); Columbia University (Other); Icahn School of Medicine at Mount Sinai (Other); Weill Medical College of Cornell University (Other); University of Pittsburgh Medical Center (Other); Methodist Health System (Other); Northwestern University (Other); NYU Langone Health (Other); University of Virginia (Other); Washington University School of Medicine (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00085148; JHUHIVDD (Other: Site Specific Identifier); 1U01AI134591-01 (NIH)
Record Dates: First submitted 2015-11-06; First posted 2015-11-11 (Estimated); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: HIV Infection
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, serum, peripheral blood mononuclear cells, tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HIV D+/R+: HIV-infected individuals who accept an organ from an HIV-infected deceased donor
  Interventions: Other: HIV-infected deceased donor organ
- HIV D-/R+: HIV-infected individuals who accept an organ from an HIV-uninfected deceased donor

INTERVENTIONS:
Other: HIV-infected deceased donor organ — HIV-infected deceased donor organ transplant
  Groups: HIV D+/R+

SUMMARY:
HIV-infected (HIV+) individuals who agree to accept and receive a solid organ transplant from an HIV+ deceased donor will be followed to determine the safety and efficacy of this practice. Some HIV+ individuals who receive a solid organ transplant from HIV-uninfected (HIV-) donors will also be followed.

DETAILED DESCRIPTION:
This is an observational study designed to evaluate safety and outcomes of solid organ transplantation in HIV+ recipients of HIV+ deceased donor organs. This study will evaluate overall survival and graft survival compared to transplantation with an HIV- organ.

In addition the study will assess potential complications of organ transplant using HIV+ deceased donors - including but not limited to - HIV superinfection, incidence and severity of graft rejection, recurrence of HIV-associated nephropathy, incidence of bacterial infections, and opportunistic infections.

ELIGIBILITY:
Inclusion Criteria:

All individuals with end-stage organ disease and HIV infection who meet standard clinical criteria for transplantation and the study inclusion and exclusion criteria will be eligible for participation in the study.

1. Participant is able to understand and provide informed consent
2. Participant meets standard listing criteria for transplant.
3. Documented HIV infection (by any licensed ELISA and confirmation by Western Blot, positive HIV Ab Immunofluorescence Assay (IFA), or documented history of detectable HIV-1 RNA).
4. Participant is > 18 years old.
5. Opportunistic Complications: None or previous history of protocol allowed opportunistic infections or neoplasms with appropriate acute and maintenance therapy and no evidence of active disease.
6. Participant CD4+ T-cell count is >/= 200/µL in the 16 weeks prior to transplant.
7. Participant most recent HIV-1 RNA < 50 copies/mL (by any FDA-approved assay performed in Clinical Laboratory Improvement Amendments (CLIA)-approved laboratory) and on a stable antiretroviral regimen. Non-consecutive viral "blips" between 50-400 copies RNA/mL will be allowed. The Federal Register HIV Organ Policy Equity (HOPE) Act Final Safeguards and Research criteria does not specify a required frequency of HIV-1 RNA monitoring to determine recipient eligibility. The most recent HIV Viral Load (VL) should be < 50 copies, but this result can be documented outside the 16 week window according to the judgement of the local clinical team and site investigator. Organ recipients who are unable to tolerate Antiretroviral Therapy (ART) due to organ failure or who have only recently started ART may have detectable viral load and still be considered eligible if the study team is confident there will be a safe, tolerable, and effective antiretroviral regimen to be used by the recipient once organ function is restored after transplantation.
8. Participant is willing to use Pneumocystis Carinii Pneumonia (PCP), herpes virus and fungal prophylaxis as indicated.

Exclusion Criteria:

1. Participant has concomitant conditions that, in the judgment of the investigators, would preclude transplantation or immunosuppression.
2. Opportunistic Complication History: Any history of progressive multifocal leukoencephalopathy (PML), chronic intestinal cryptosporidiosis of > 1 month duration, or primary Central Nervous System (CNS) lymphoma.
3. Participant has a history of any neoplasm except for the following: resolved Kaposi's sarcoma, in situ anogenital carcinoma, adequately treated basal or squamous cell carcinoma of the skin, solid tumors (except primary CNS lymphoma) treated with curative therapy and disease free for more than 5 years. History of renal cell carcinoma requires disease free state for 2 years. History of leukemia and disease-free duration will be per site policy.
4. Participant is pregnant or breastfeeding. Note: Participants who become pregnant post-transplant will continue to be followed in the study and will be managed per clinical practice. Women that become pregnant should not breastfeed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All individuals with end-stage organ disease and HIV infection who meet standard clinical criteria for transplantation and the study inclusion and exclusion criteria will be eligible for participation in the study.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2020-06-12 (Actual); Study Completion 2023-06-16 (Actual)

PRIMARY OUTCOMES:
Survival | One year
  Patient survival at one year

SECONDARY OUTCOMES:
Graft survival | one year, two years, 3 years, 4 years
  Transplanted organ function
Graft rejection | One year
  Incidence and severity of organ rejection
HIV disease progression | through study completion, up to 4 years
  Incidence of virologic breakthrough or failure
Antiretroviral resistance and X4 tropic virus | through study completion, up to 4 years
  incidence of new antiretroviral drug resistance and/or X4 tropic virus
Incidence of bacterial, fungal, viral, and other opportunistic infection | through study completion, up to 4 years
  incidence of bacterial, fungal, viral, and other opportunistic infections
Surgical complications | within the first 3 months
  incidence of surgical and vascular transplant complications
Recurrent HIV-associated nephropathy | through study completion, up to 4 years
  incidence of recurrent HIV-associated nephropathy in kidney recipients
Incidence of post-transplant Malignancy | through study completion, up to 4 years
  incidence of post-transplant malignancies
Incidence of HIV superinfection in blood and/or tissue | measured at 3 months, 6 months, year 1, year 2, year 3, year 4
  Incidence of HIV superinfection in blood and/or tissue
HIV latent reservoir | measured at 3 months, 6 months, year 1, year 2, year 3, year 4
  Frequency of infected CD4 T cells in blood
Immune activation | measured at 3 months, 6 months, year 1, year 2, year 3, year 4
  Cytokine levels

CONTACTS AND LOCATIONS:
Overall Officials: Christine Durand, MD, Principal Investigator — Johns Hopkins University
Locations (18):
- United States (18):
  - University of Colorado Denver, Aurora, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Illinois at Chicago, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Maryland, Institute of Human Virology, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - Washington University School of Medicine, St Louis, Missouri
  - New York University School of Medicine, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Columbia University Medical Center, New York, New York
  - Weill Cornell Medical College, New York, New York
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Methodist Health System, Dallas, Texas
  - University of Virginia, Charlottesville, Virginia

REFERENCES:
- [Derived] Arant EC, Davy-Mendez T, Liang T, Rodrigues M, Gay CL, Rana MM, Friedman-Moraco R, Gilbert A, Stock P, Mehta SA, Mehta S, Stosor V, Pereira MR, Morris MI, Hand J, Aslam S, Malinis M, Haidar G, Small CB, Santos CAQ, Schaenman J, Baddley JW, Wojciechowski D, Blumberg EA, Ranganna K, Adebiyi O, Elias N, Castillo-Lugo JA, Giorgakis E, Apewokin S, Morsheimer M, van Delden C, Manuel O, Mueller NJ, Neofyotos D, Tobian AAR, Massie A, Segev DL, Werbel W, Durand CM. Infections After Kidney Transplantation From Donors With Human Immunodeficiency Virus (HIV) to Recipients With HIV. Clin Infect Dis. 2026 Jan 12:ciaf656. doi: 10.1093/cid/ciaf656. Online ahead of print. PMID 41524130
- [Derived] Benner SE, Zhu X, Hussain S, Florman S, Eby Y, Fernandez RE, Ostrander D, Rana M, Ottmann S, Hand J, Price JC, Pereira MR, Wojciechowski D, Simkins J, Stosor V, Mehta SA, Aslam S, Malinis M, Haidar G, Massie A, Smith ML, Odim J, Morsheimer M, Quinn TC, Laird GM, Siliciano R, Balagopal A, Segev DL, Durand CM, Redd AD, Tobian AAR. HIV-Positive Liver Transplant Does not Alter the Latent Viral Reservoir in Recipients With Antiretroviral Therapy-Suppressed HIV. J Infect Dis. 2023 Nov 2;228(9):1274-1279. doi: 10.1093/infdis/jiad241. PMID 37379584
- [Derived] Werbel WA, Brown DM, Kusemiju OT, Doby BL, Seaman SM, Redd AD, Eby Y, Fernandez RE, Desai NM, Miller J, Bismut GA, Kirby CS, Schmidt HA, Clarke WA, Seisa M, Petropoulos CJ, Quinn TC, Florman SS, Huprikar S, Rana MM, Friedman-Moraco RJ, Mehta AK, Stock PG, Price JC, Stosor V, Mehta SG, Gilbert AJ, Elias N, Morris MI, Mehta SA, Small CB, Haidar G, Malinis M, Husson JS, Pereira MR, Gupta G, Hand J, Kirchner VA, Agarwal A, Aslam S, Blumberg EA, Wolfe CR, Myer K, Wood RP, Neidlinger N, Strell S, Shuck M, Wilkins H, Wadsworth M, Motter JD, Odim J, Segev DL, Durand CM, Tobian AAR; HOPE in Action Investigators. National Landscape of Human Immunodeficiency Virus-Positive Deceased Organ Donors in the United States. Clin Infect Dis. 2022 Jun 10;74(11):2010-2019. doi: 10.1093/cid/ciab743. PMID 34453519
- [Derived] Bonny TS, Kirby C, Martens C, Rose R, Desai N, Seisa M, Petropoulos C, Florman S, Friedman-Moraco RJ, Turgeon NA, Brown D, Segev DL, Durand CM, Tobian AAR, Redd AD. Outcomes of donor-derived superinfection screening in HIV-positive to HIV-positive kidney and liver transplantation: a multicentre, prospective, observational study. Lancet HIV. 2020 Sep;7(9):e611-e619. doi: 10.1016/S2352-3018(20)30200-9. Epub 2020 Jul 27. PMID 32730756